CLINICAL TRIAL: NCT04424212
Title: CoronaCope - Internet-based Cognitive Behavioural Therapy for Adults Suffering From Mental Health Problems Related to the Coronavirus Pandemic
Brief Title: ICBT for Mental Health Problems Related to the Coronavirus Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoronaCope
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Depression and Quality of Life Related to the Coronavirus Pandemic
Keywords: Corona; COVID-19; Internet-delivered cognitive-behavioral therapy (ICBT); Depression; Quality of life
MeSH Terms: conditions — Depression; COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either control or intervention group. Participants in the control group will receive the same treatment once the intervention group has finished the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group CoronaCope (Experimental): ICBT, were participants receive 8 out of 15 possible modules depending on their current problems and needs, 7 week long internet intervention for reducing mental health issues related to the coronavirus pandemic.
  Interventions: Behavioral: Intervention group CoronaCope
- Control group (No Intervention): Participants in the control group will be instructed to wait. Once intervention group will be finished, participants in control group will be able to access the same intervention.

INTERVENTIONS:
Behavioral: Intervention group CoronaCope — Intervention based on cognitive behavioural therapy principles and adapted to the coronavirus pandemic situation. Intervention's main purpose is to mental health issues such as depressive symtoms, stress, worry and anxiety related to the coronavirus pandemic and increase quality of life in the current situation. Intervention contains psycho-educational elements as well as examples and exercises.
  Arms: Experimental: Intervention group CoronaCope

SUMMARY:
The study seeks to investigate the effects of a guided internet-based cognitive behavioral therapy (ICBT) programme a on adult mental health problems related to the current coronavirus pandemic. ICBT will be compared to a wait-list control group.

Participants will be recruited in Sweden with a nationwide recruitment.

DETAILED DESCRIPTION:
The study is set up as a randomized controlled trial. Quality of life, depressive symptoms, anxiety, sleep problems and traumatic stress will be measured. Given uncertainties regarding the psychological effects of Covid-19 pandemic a transproblematic tailored treatment approach will be used that has been tested in several previous trials. However, the present program has been adapted for the target population of people who are affected by the societal and individual consequences of the pandemic. The study does not focus on people who have or have had the corona virus.

ELIGIBILITY:
Inclusion Criteria:

* Experience mental health problems that are caused or exacerbated by the corona pandemic and/or its consequences
* 18 years or older.
* Adequate ability to understand and speak Swedish.
* Access to the internet and a smartphone/computer.

Exclusion Criteria:

* Other ongoing psychological treatment or counselling that interfere with trial treatment.
* Recent (within the past 3 months) changes in the dose of psychotropic medication.
* Any severe psychiatric or somatic conditions that would interfere with trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Becks Depression Inventory-II | Change between baseline and end of treatment after seven weeks.
  Measure of depressive symptoms. Possible range for the total sum: 0 to 63 (created by summing up the score from each item) with a higher score indicating a higher level of depressive symptoms. Clinical ranges for minimal, mild, moderate and severe major depressive disorder are considered to be 0-13, 13-19, 20-28, and 29-63 points.
Brunnsviken Brief Quality of Life Scale | Change between baseline and end of treatment after seven weeks.
  Measure of quality of life, total score ranging from 0 to 96 with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.

SECONDARY OUTCOMES:
Patient Health Questionnaire | Change between baseline and end of treatment after seven weeks.
  Measure of depressive symptoms. Possible range for the total sum: 0 to 27 (created by summing up the score from each item) with a higher score indicating higher levels of depression. Clinical cut-offs for mild, moderate, moderately severe and severe major depressive disorder are considered to be 5, 10, 15, and 20 points.
Alcohol Use Disorder Identification Test | Change between baseline and end of treatment after seven weeks.
  The Alcohol Use Disorders Identification Test is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. 10 items and scores ranging from 0-40 with higher scores indicating a higher level of alcohol use.
Insomnia Severity Index | Change between baseline and end of treatment after seven weeks.
  Measure of insomnia severity and symptoms of disordered sleep. The total score can range between 0 (no sleep problems) to 28 (severe sleep problems and insomnia) with higher scores indicating severer levels of sleeping problems. Norm score ranges include low likelihood of sleep problems (0 to 7 points), some sleep problems (8 to 14 points), moderate sleep problems (15 to 21 points), severe sleep problems (22 to 28 points).
The CoRonavIruS Health Impact Survey | At baseline
  Screening for health impact and exposure of the coronavirus pandemic, with higher scores indicating a more severe impact from the coronavirus pandemic.
Impact of Event Scale-Revised | Change between baseline and end of treatment after seven weeks.
  Assesses subjective distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The Impact of Event Scale-Revised yields a total score (ranging from 0 to 88) with a higher score indicate more severe distress caused by the traumatic events.
Perceived Stress Scale | Change between baseline and end of treatment after seven weeks.
  It is a measure of the degree to which situations in one's life are appraised as stressful. It contains 10 items that are scored on a range between 0 (never) to 4 (very often). The total score can range from 0-56 and a higher score reflects higher levels of perceived stress.
Becks Depression Inventory-II | Change between posttreatment and 12-month follow-up.
  Same as during the treatment phase.
Brunnsviken Brief Quality of Life Scale | Change between posttreatment and 12-month follow-up.
  Same as during the treatment phase.
Dimensions of Anger Reactions (DAR-5) Questionnaire | Change between posttreatment and 12-month follow-up.
  The DAR-5 measures anger and its frequency, intensity, duration, level of aggression and impact on functioning during the last 4 weeks. The total severity score range between 5-25. Higher scores indicate that you are experiencing psychological distress and functional impairment as a result of your anger.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden